CLINICAL TRIAL: NCT03993561
Title: Survivorship After Head And Neck Cancer: Validation of Treatment Summary and Survivorship Care Plans
Brief Title: Treatment Summary and Survivorship Care Plans (TSSP)
Acronym: SHARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Danielle MacNeil, Assistant Professor - Department of Otolaryngology Head & Neck Surgery, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 114194
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Survivorship; Head and Neck Cancer
Keywords: treatment summary and survivorship care plan; intervention; head and neck cancer survivors
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective, pilot trial at a single centre with 1 group of 20 adults. The study group will receive a one-hour treatment summary and survivorship care plan (TSSP) intervention specifically tailored to the needs of head and neck cancer patients based on the best available evidence and consultation with patients and a multidisciplinary team of head and neck cancer specialists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TSSP Group (Experimental): A one-hour treatment summary and survivorship care plan (TSSP) intervention specifically tailored to the needs of head and neck cancer patients based on the best available evidence and consultation with patients and a multidisciplinary team of head and neck cancer specialists will be provided
  Interventions: Other: Treatment summary and survivorship care plan

INTERVENTIONS:
Other: Treatment summary and survivorship care plan — Individually tailored counselling session will be implemented within 1 month of treatment completion.

SUMMARY:
The aim of the study is to establish the highest level of evidence to evaluate treatment summary and survivorship care plans (TSSPs) by piloting the TSSPs on patients with HNC.

Hypothesis: HNC patients who receive the intervention of the TSSP will have an increased rate of implementation of recommendations for their needs, greater adherence with follow-up schedules, improved quality of life and improved satisfaction with post-treatment care.

Aim 1 (Validation of TSSP): To validate a treatment summary and survivorship care plan (TSSP) intervention specifically tailored to the needs of HNC patients based on the best available evidence.

Approach: In the first phase of the project the investigators will pilot the London Heath Sciences Centre TSSP with head and neck cancer survivors and then have the TSSP extensively reviewed and modified by our multidisciplinary head and neck oncology treatment team.

Aim 2 (Evaluation of TSSP): To evaluate the implementation of a TSSP in survivors of head and neck cancer compared to usual treatment in a randomized fashion to determine whether TSSPs result in improved implementation of recommendations for HNC survivors and improved quality of life and satisfaction.

Approach: In the second phase of the project the investigators will conduct a randomized controlled trial to compare patient reported outcomes in HNC patients who have received the TSSP to patients who have not received the TSSP.

DETAILED DESCRIPTION:
Validation of TSSP: The investigators have performed an extensive literature review to create a comprehensive draft TSSP specifically tailored for HNC patients. The investigators will pilot this study among 20 head and neck cancer survivors. Once the investigators have the feedback from the pilot patients, the investigators will conduct a focus group with the members of our head and neck multidisciplinary group to gain input on the TSSP.

Evaluation of TSSP: The investigators will recruit head and neck cancer survivors with curable stage I-IVA head and neck mucosal cancer at a tertiary level cancer center in Ontario. Patients will receive a survivorship care plan (TSSPs) intervention. The intervention will consist of a survivorship care nurse or radiation therapist counseling session coupled with the provision of individualized TSSPs to patients and their health care providers. After a baseline telephone or in-person interview, eligible participants will be provide with the TSSP.

The primary outcome will be physician implementation of TSSP care recommendations over the course of 12 months, assessed by quarterly patient interviews. Secondary outcomes will include adherence to recommended follow-up schedules, quality of life using validated measures and patient satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* willing to provide informed consent
* diagnosis of stage I-IVA head and neck mucosal cancer (larynx, hypopharynx, oral cavity, oropharynx, nasopharynx)
* last definitive treatment (surgery, chemotherapy, radiotherapy) at least 1 month but no greater than 3 months from enrollment
* English speaking

Exclusion Criteria:

* Second concurrent non-cutaneous malignancy
* metastatic disease
* clinically apparent cognitive impairment
* unable or unwilling to complete questionnaires
* suspected residual disease after treatment completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Physician implementation of TSSP | 12 months
  Physician implementation of treatment summaries and survivorship care plans (TSSP) recommendations over the course of 12 months, assessed by quarterly patient interviews.

SECONDARY OUTCOMES:
Satisfaction with Care and Communication | baseline and 12 months post-treatment
  8-item questionnaire measuring patient level of satisfaction with follow-up care since head and neck cancer treatment ended; 4 questions are ranked using a 6-point Likert scale (1 = Never and 6 = Always), 1 item uses a 5-point likert scale (1 = Definitely yes; 5 = Definitely not); 2 items use a scale of 0-10 (0 = not at all satisfied and 10 = very satisfied); and one item utilized a Yes or No response format. Total scores range from 5 to 50;
Patient Self-Efficacy (PEPPI) | baseline and 12 months post-treatment
  Five item patient self-efficacy measured on a scale of 0 to 10 (0 = not confident at all, 10 = extremely confident); higher scores indicate better satisfaction with care; Total scores range from 0 to 50;
KATZ Comorbidity Scale | baseline and 12 months post-treatment
  Patient rated comorbidity scale based on the Charlson Comborbidity index. Thirty-five item scale measures the presence or absence of different health conditions. Each item utilizes a Yes/No format; Yes' are given a point of 1 and No's are scored 0; Higher scores indicate the presence of a greater number of co-morbidities and lower scores; Total scores range from 0 to 35;
36-Item Short Form Survey Instrument (SF-36) | baseline and 12 months post-treatment
  36 item scale to measure patient health and wellbeing from the patient perspective; Eight subscale scores are generated for the following domains: 1) physical functioning, 2) role-physical, 3) bodily pain, 4) general health, 5) vitality, 6) social functioning, 7) role-emotional, and 8) mental health; Item scales range from 3 to 6 point Likert scales and Yes/No response formats; items are recoded to a scale of 0 to 100; after recoding, averages for each subscale are calculated so that each subscale has a range of 0 to 100 (0 being poor functioning and 100 excellent functioning); higher subscale scores indicate better health.
Personal Health Questionnaire Depression Scale (PHQ-8) | baseline and 12 months post-treatment
  Eight-item self-reported depression scale; each item is scored using a 4-point likert scale (0 = Not at all, 3 = Nearly every day); Total scores range from 0 to 24; A score of 10 or greater is considered major depression, 20 or more is severe depression;
Knowledge and Preparedness for Survivorship Scale (PLANS scale) | baseline and 12 months post-treatment
  Sixteen- item knowledge of survivorship issues questionnaire; Items 1-11 use a 4-point scale (1 = Strongly disagree; 4 = Strongly agree) and addresses knowledge of survivorship issues; items 12 to 16 utilize a 10-point scale (1 = Not at all confident; 10 = Extremely Confident) and evaluate patient preparedness for survivorship; Subscale total scores for Knowledge of Survivorship Issues subcale range from 11 to 44 with higher scores indicating better knowledge of survivorship issues; The Preparedness for Survivorship (items 12-16) subscale score ranges from 5 to 50 with higher scores indicating greater level of confidence regarding preparedness for survivorship
Short-Form Patient Satisfaction Questionnaire (PSQ-18) | baseline and 12 months post-treatment
  Eighteen-item patient satisfaction with care questionnaire using a 5-point Likert scale (1 = Strongly agree; 5 = Strongly disagree); Five subscale scores are generated by calculating averages of items that belong to that particular subscale: General Satisfaction, Technical Quality, Interpersonal Manner, Communication, Financial Aspects, Time Spent with Doctor, Accessibility and Convenience; Each subscale score ranges from 1 to 5 with higher scores reflecting greater level of satisfaction with care;
Social support survey | baseline and 12 months post-treatment
  Nineteen-item scale measuring social, tangible and emotional support; Each item is ranked on a 5-point likert scale (1 = None of the time and 5 = All of the time); Higher scores indicate greater social support;

CONTACTS AND LOCATIONS:
Overall Officials: Danielle MacNeil, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon request